CLINICAL TRIAL: NCT00531089
Title: A Phase II Study Evaluating the Efficacy of Rituximab in the Management of Patients With Relapsed/Refractory Thrombotic Thrombocytopenic Purpura (TTP) - Hemolytic Uremic Syndrome (HUS)
Brief Title: Rituximab in Patients With Relapsed or Refractory TTP-HUS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Apheresis Group (Other); Hoffmann-La Roche (Industry); McMaster University (Other)
Responsible Party: Canadian Apheresis Group, Canadian Apheresis Group
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAG-1
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2007-09

CONDITIONS: Thrombotic Thrombocytopenic Purpura; Hemolytic Uremic Syndrome
Keywords: TTP; thrombotic thrombocytopenic purpura; HUS; hemolytic uremic syndrome; plasma exchange
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic; Hemolytic-Uremic Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study group (Experimental): All patients in the study will be in the study group and will receive rituximab. There is no "control" arm.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab will be administered on weeks 1, 2, 3, and 4 at a dose of 375 mg/m2 per infusion. Premedications (prednisone 50 mg, diphenhydramine 50 mg, acetaminophen) will be administered prior to study infusion. Patients will also be treated with plasma exchange as per institution/apheresis centre.
  Other Names: Rituxan, rituximab

SUMMARY:
The general objective of this study is to assess the efficacy and safety of Rituximab in the management of patients with refractory or relapsed thrombotic thrombocytopenic purpura-hemolytic uremic syndrome (TTP-HUS). There have been several case reports and case series describing the use of Rituximab in patients with TTP-HUS; however its use has not been studied in a large trial. It is hypothesized that Rituximab may ameliorate the severity of certain cases of TTP-HUS by decreasing the number of activity of B-cells which may result in decreased production of the ADAMTS13 protease inhibitor. Patients with TTP-HUS not responding to standard therapy or patients with relapsed disease may have particular benefit. Treatments that decrease the frequency of relapse or shorten the time to remission of TTP-HUS will be of benefit by decreasing the need for blood product support.

ELIGIBILITY:
Inclusion Criteria:

* any patient 18 years or older diagnosed with relapsed or refractory TTP-HUS requiring therapy

Exclusion Criteria:

* alternate cause of hemolytic microangiopathy (evidence of DIC, malignant hypertension, vasculitis, anti-phospholipid antibody syndrome, post-partum acute renal failure)
* congenital or familial TTP
* TTP occuring post-stem cell, bone marrow, or solid organ transplant
* drug-induced TTP
* pregnancy or breast-feeding
* history of hepatitis B or C infection
* prior rituximab treatment
* active or metastatic cancer
* other causes of thrombocytopenia such as ITP, myelodysplastic syndrome, confirmed or suspected drug-induced thrombocytopenia
* refusal to receive blood products
* hypersensitivity to blood products, plasma products, murine proteins, or any component of the Rituximab formulation
* geographic inaccessibility
* co-morbid illness limiting life expectancy to less than 2 months independent of TTP
* failure to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving all: (1) platelet count >150x109/L; (2) LDH < 1.5 x normal; (3) no requirement for plasma exchange therapy; (4) asymptomatic. | 8 weeks after initiation of therapy

SECONDARY OUTCOMES:
proportion of patients with platelet count greater than 150 x 109/L | 8 weeks
proportion of patients with LDH < 1.5 X normal | 8 weeks
proportion of patients with no requirement for plasma exchange therapy | 8 weeks
proportion of patients who are asymptomatic (no new neurological symptoms ans stabilization of previous neurological symptoms | 8 weeks
clinical response (CR, PR, non-response) | 52 weeks
frequency of relapse | 52 weeks
mortality | 52 weeks
changes from baseline in platelet counts, LDH, ADAMTS13 protease level, ADAMTS13 inhibitor level | 8, 12, 24, 52 weeks
toxicity and clinical safety as assessed by monitoring of adverse events, laboratory parameters, vital signs during infusion, and immediate tolerability | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Webert, E, Principal Investigator — Hamilton Health Sciences Corporation; Ronan Foley, MD, Principal Investigator — Hamilton Health Sciences Corporation; Gail Rock, MD, Study Director — Canadian Apheresis Group; William Clark, MD, Study Director — University of Western Ontario/London Health Sciences; David Barth, MD, Study Director — University of Toronto
Locations (11):
- Canada (11):
  - Foothills Medical Centre, Calgary Health REgion Apheresis Service, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Winnipeg Regional Health Authority, Apheresis Department, Winnipeg, Manitoba
  - St. John Regional Hospital, Saint John, New Brunswick
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, Westminister Campus, London, Ontario
  - Princess Margaret Hospital, ABMT/Apheresis Unit, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - St. Paul's Hospital Apheresis Unit, Saskatoon, Saskatchewan